CLINICAL TRIAL: NCT03051906
Title: Anti PD-L1 Durvalumab Combined With Cetuximab and Radiotherapy in Locally Advanced Squamous Cell Carcinoma of the Head and Neck: a Phase I/II Study
Brief Title: Durvalumab, Cetuximab and Radiotherapy in Head Neck Cancer
Acronym: DUCRO-HN
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Professor; Chair of Radiation Oncology Department, Azienda Ospedaliero-Universitaria Careggi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DUCRO-HN; 2016-004668-20 (EudraCT Number)
Record Dates: First submitted 2017-02-06; First posted 2017-02-14 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Head and Neck Neoplasms
Keywords: Carcinoma, squamous cell; Head and Neck Neoplasms; Radiotherapy; Immunotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — durvalumab; Cetuximab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Durvalumab, Cetuximab and Radiotherapy followed by adjuvant Durvalumab (6 months)
  Interventions: Biological: Durvalumab; Biological: Cetuximab; Radiation: Intensity modulated radiation therapy (IMRT)

INTERVENTIONS:
Biological: Durvalumab — Durvalumab given intravenously at 1500 mg every 4 weeks; first two cycles concurrent with RT + cetuximab, 6 cycles after the end of RT as adjuvant treatment; treatment will be continued for a maximum of 8 months (concurrent phase included).
Biological: Cetuximab — Cetuximab given intravenously weekly at 400mg/m2 loading dose 1 week before RT start, then 250 mg/m2 weekly thereafter.
Radiation: Intensity modulated radiation therapy (IMRT) — A total dose of 69.9 Gy will be given with 2.12 Gy dose per fraction, delivered in 33 fractions over 7 weeks.

SUMMARY:
In over 60% of cases, squamous cell carcinoma of the head and neck (SCCHN) is discovered at a loco-regionally advanced stage that requires a combined multimodal strategy in order to pursue a curative intent. Bonner et al demonstrated that the combination of radiation (RT) with Cetuximab (CTX), a chimeric mouse IgG1 monoclonal anti-EGFR antibody, results in better median locoregional control and overall survival compared with RT alone without an increased rate of > G3 acute toxicity or detrimental effect on compliance and quality of life. However, subsequent negative trials (RTOG 0522) led to the hypothesis that in unselected patient populations the benefit of CTX may be diluted due to the molecular heterogeneity of SSCHN. Moreover, the absence of biomarkers predictive of response to anti-EGFR treatment may in part be explained by the observation that other factors play a role in favoring its anticancer effect, namely immunologic mechanisms. It has been demonstrated that SCCHN is an immunosuppressive disease characterized by prominent immuno-escape mechanisms, such as induction of a tumor-permissive cytokine profile and qualitative/quantitative lymphocyte deficiencies, occurrence of anergy in major immune effector cells and poor antigen presentation. Given these observations, it has been postulated that SCCHN may benefit from immunotherapeutic strategies, primarily aimed at PD-L1/PD1 checkpoint blockade. Segal et al (Asco 2015) reported preliminary results on the use of Durvalumab in pretreated patients with recurrent/metastatic SCCHN. Durvalumab is a humanized monoclonal IgG1 antibody that blocks PD-L1 binding to PD-1 and CD80 with high affinity and selectivity, thereby promoting activity of tumor-specific effector T cells and global anti-tumor immune response. Out of 64 treated patients, 51 patients were available for the preliminary efficacy analysis: promisingly, the overall response rate was 12% (25% in PD-L1 positive patients). To date, no clinical trial, specifically designed for SCCHN, testing PD-L1 targeted agents has been completed, nor have been initiated combination strategies of CTX, RT and PD1/PD-L1 antibodies in the curative setting. Taken all data together, a strong rationale may support the combination of Durvalumab, anti-EGFR therapy such as CTX and RT in order to revert the SCCHN-induced immune suppression and maximize treatment efficacy, ultimately through enhanced, CTX-mediated immune mechanisms and maximized RT-specific cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization obtained from the patients prior to performing any protocol-related procedures, including screening evaluations
* Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma (including the histological variants papillary squamous cell carcinoma and basaloid squamous cell carcinoma) of the oropharynx, hypopharynx and larynx
* For patients with oropharyngeal cancer only: confirmed HPV status by HPV- DNA ISH prior to registration
* Confirmed PD-L1-positive or -negative status by the Ventana SP263 IHC assay
* Patients agree to provide their smoking history prior to registration
* Clinical stage of HPV-negative oropharynx and all hypopharynx and larynx: T1-2, N2a-N3 or T3-4, any N (AJCC 7th ed.), including no distant metastases
* Clinical stage of HPV-positive oropharynx: T2-4, N2b-N3 (AJCC 7th ed.), including no distant metastases with smoking history ≥ 10 pack/years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow: absolute neutrophil count ≥ 1,500/μl, platelets ≥ 100,000/μl, hemoglobin ≥ 9 g/dL
* Adequate hepatic function: total bilirubin ≤ 1.5 X upper normal limit (UNL), aspartate aminotransferase (AST) ≤ 2.5 X UNL, alanine aminotransferase (ALT) ≤ 2.5 X UNL
* Adequate renal function: calculated serum creatinine clearance >40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection

Exclusion Criteria:

* Histologically confirmed head and neck cancer of any other primary anatomic location in the head and neck not specified in the inclusion criteria including patients with SCCHN of unknown primary or non-squamous histologies (eg, nasopharynx or salivary gland)
* Clinical stage of HPV-negative oropharynx and all hypopharynx and larynx: T1-2, N0-1 (AJCC 7th ed.)
* Clinical stage of HPV-positive oropharynx: T1-2, N0-N2a (AJCC, 7th ed.) or any T, any N with smoking history of < 10 pack/years
* History of another primary malignancy except for: malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; adequately treated carcinoma in situ without evidence of disease (eg, carcinoma in situ of the breast, oral cavity and cervix are all permissible); low risk prostate cancer based on NCCN criteria on active surveillance, not candidate to any curative treatment given the extremely low likelihood of disease progression
* Gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Prior use of cetuximab or other anti-EGFR therapy
* Any previous treatment with PD-1 or PD-L1 inhibitors, including Durvalumab
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of Durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity (>CTCAE grade 2) from previous anti-cancer therapy
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
* Active or prior documented autoimmune disease within the past 2 years (subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment within the past 2 years are not excluded)
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Severe, active co-morbidity, defined as follows:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
* Transmural myocardial infarction within the last 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* Known history of active infection including tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of the experimental regimen (Durvalumab, Cetuximab and Radiotherapy) | 2-year PFS
  Progression-free survival according to Recist 1.1

SECONDARY OUTCOMES:
To assess the number of participants with treatment-related adverse events according to CTCAE v.4 | Within 90 days of end of treatment (last infusion of Durvalumab scheduled at 29th week; EoT)
  Acute toxicity according to CTCAE v. 4
To assess the tolerability of the experimental regimen (Durvalumab, Cetuximab and Radiotherapy) | Within 90 days of end of treatment (last infusion of Durvalumab scheduled at 29th week; EoT)
  Relative dose intensity (RDI) of Durvalumab, Cetuximab and Radiotherapy
To assess the efficacy of the experimental regimen (Durvalumab, Cetuximab and Radiotherapy) | 2-year LRC
  Locoregional control (LRC) according to Recist 1.1
To assess the efficacy of the experimental regimen (Durvalumab, Cetuximab and Radiotherapy) | 2-year OS
  Overall Survival (OS) according to Recist 1.1
To assess the efficacy of the experimental regimen (Durvalumab, Cetuximab and Radiotherapy) | 5-year OS
  Overall Survival (OS) according to Recist 1.1
To assess the number of participants with treatment-related adverse events | Beyond 90 days of end of treatment (last infusion of Durvalumab scheduled at 29th week; EoT)
  Late toxicity according to CTCAE v.4
To assess health-related quality of life (HRQoL) in patients treated with the experimental regimen (Durvalumab, Cetuximab and Radiotherapy) | Baseline, within 2 weeks of end of treatment (EoT), 12 months (change over time)
  EORTC-QLQ C30, EORTC-QLQ H&N35 questionnaires

IPD SHARING:
Plan to Share IPD: Yes
Clinical and biologic (translational) individual data will be available after the end of study

REFERENCES:
- [Derived] Bonomo P, Desideri I, Mangoni M, Saieva C, Loi M, Becherini C, Cerbai C, Ganovelli M, Salvestrini V, Stocchi G, Zani M, Palomba A, Livi L. Durvalumab with cetuximab and radiotherapy for locally advanced squamous cell carcinoma of the head and neck: A phase 1/2 trial. Radiother Oncol. 2022 Apr;169:64-70. doi: 10.1016/j.radonc.2022.02.008. Epub 2022 Feb 11. PMID 35157978
- [Derived] Bonomo P, Desideri I, Loi M, Mangoni M, Sottili M, Marrazzo L, Talamonti C, Greto D, Pallotta S, Livi L. Anti PD-L1 DUrvalumab combined with Cetuximab and RadiOtherapy in locally advanced squamous cell carcinoma of the head and neck: A phase I/II study (DUCRO). Clin Transl Radiat Oncol. 2018 Feb 7;9:42-47. doi: 10.1016/j.ctro.2018.01.005. eCollection 2018 Feb. PMID 29594250